CLINICAL TRIAL: NCT02429258
Title: Effect of Dapagliflozin on 24-hour Blood Glucose in T2DM Patients Inadequately Controlled With Either Metformin Or Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1690L00026
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Farxiga with metformin or insulin (Experimental): Farxiga with metformin (>/=1500mg/day) or insulin (>/=30 units/day) and up to 2 OAD medications
  Interventions: Drug: Farxiga; Drug: Metformin; Drug: Insulin
- Placebo with metformin or insulin (Placebo Comparator): Placebo with metformin (>/=1500mg/day) or insulin (>/=30 units/day) and up to 2 OAD medications
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Insulin

INTERVENTIONS:
Drug: Farxiga — Farxiga 10mg/day
  Arms: Farxiga with metformin or insulin
Drug: Placebo — Placebo
  Arms: Placebo with metformin or insulin
Drug: Metformin — Metformin background therapy >/= 1500mg/day
Drug: Insulin — Insulin >/= 30 units

SUMMARY:
Effect of Dapagliflozin on 24-hour Blood Glucose in Type 2 Diabetes Patients Inadequately Controlled With Either Metformin Or Insulin

DETAILED DESCRIPTION:
Effect of Dapagliflozin on 24-hour Blood Glucose in 92 Type 2 Diabetes Patients Inadequately Controlled With Either Metformin Or Insulin

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM)
* Treated with either stable dose of metformin alone > or = to 1500mg/day or stable dose of insulin > or = to 30 units/day and up to 2 OAD medications for at least 8 weeks
* Hemoglobin A1c (HbA1c) 7.5% to 10.5% at screening
* Body mass index (BMI) < or = to 45 kg/m2

Exclusion Criteria:

* For patients who enter the study taking a stable dose of metformin, history of taking OAD medications other than metformin during the 8 weeks prior to screening or have been on insulin therapy within 1 year of screening
* For patients who enter the study taking insulin, history of taking any other therapy outside of the stable insulin and up to 2 OAD medications for 8 weeks prior to screening.
* Use of sulfonylureas during the 8 weeks prior to screening
* Prior exposure to dapagliflozin or any sodium-glucose co-transporter 2 (SGLT-2) inhibitor
* Ingestion of any medication know to affect glucose metabolism for >7 consecutive days during the 3 months prior to screening
* Ingestion of prescription or over the counter weight loss medication during 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Huntington Park, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, West Hills, California
  - Research Site, Cooper City, Florida
  - Research Site, Miami, Florida
  - Research Site, Evanston, Illinois
  - Research Site, Oxon Hill, Maryland
  - Research Site, Henderson, Nebraska
  - Research Site, Brooklyn, New York
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Franklin, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Bartlett, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Hurst, Texas
  - Research Site, Renton, Washington

REFERENCES:
- [Derived] Henry RR, Strange P, Zhou R, Pettus J, Shi L, Zhuplatov SB, Mansfield T, Klein D, Katz A. Effects of Dapagliflozin on 24-Hour Glycemic Control in Patients with Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Technol Ther. 2018 Nov;20(11):715-724. doi: 10.1089/dia.2018.0052. Epub 2018 Sep 14. PMID 30222367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 226 subjects signed the informed consent form (ICF), and 132 subjects were screened to randomize a total of 100 subjects.
Groups:
- Dapagliflozin: Dapagliflozin + Metformin or Insulin
- Placebo: Placebo + Metformin or Insulin
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 50 | 50
Completed | 48 | 49
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: 100 subjects were included in the safety and ITT population. 99 subjects were included in the evaluable population. 1 subject did not meet the I/E criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (7.11) | 56.8 (9.71) | 56.9 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 26 | 25 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 11 | 14 | 25
  White | 39 | 36 | 75
  American Indian and Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Other | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (5.92) | 33.2 (5.59) | 33.8 (5.75)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage] | 8.31 (0.785) | 8.37 (0.810) | 8.34 (0.794)

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Mean Weighted Glucose (MWG) From Baseline to End of Treatment (Week 4) Using the Continuous Glucose Monitoring (CGM) System
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mg/dL | -18.2 (4.33) | 5.8 (4.25)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -24.0, 95% CI [-36.1 to -12.0], Standard Error of Mean 6.08

2. Secondary Outcome: Change in the 24-hour Mean Ampitude of Glucose Excursions (MAGE) From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mg/dL | -10.0 (4.14) | 5.3 (4.06)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Final Values) = -15.3, 95% CI [-26.8 to -3.8], Standard Error of Mean 5.80

3. Secondary Outcome: Change in Percentage of CGM Readings Over 24-hours With Plasma Glucose <70 mg/dL From Baseline to Week 4 - ITT Population
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: Change in percentage
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
Change in percentage | 0.3 (0.30) | -0.6 (0.29)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.023, ANCOVA; Mean Difference (Final Values) = 1.0, 95% CI [0.1 to 1.8], Standard Error of Mean 0.42

4. Secondary Outcome: Change in Percentage of CGM Readings Over 24-hours With Plasma Glucose Between 70 mg/dL and 180 mg/dL From Baseline to Week 4 - ITT Population
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: Change in percentage
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
Change in percentage | 12.2 (2.60) | -2.8 (2.55)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 15.0, 95% CI [7.7 to 22.2], Standard Error of Mean 3.65

5. Secondary Outcome: Change in Percentage of CGM Readings Over 24-hours With Plasma Glucose >180 mg/dL From Baseline to Week 4 - ITT Population
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: Change in percentage
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
Change in percentage | -12.6 (2.65) | 3.5 (2.60)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -16.1, 95% CI [-23.5 to -8.7], Standard Error of Mean 3.72

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mg/dL | -26.2 (5.99) | 3.6 (5.98)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -29.7, 95% CI [-46.6 to -12.9], Standard Error of Mean 8.47

7. Secondary Outcome: Change in 4-hour Mean Weighted Post-prandial Glucose (PPG) (After the Standardized Breakfast Meal) From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mg/dL | -50.9 (6.54) | -10.0 (6.39)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -40.8, 95% CI [-59.0 to -22.7], Standard Error of Mean 9.14

8. Secondary Outcome: Change in HbA1c From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: % Alc
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
% Alc | -0.51 (0.07) | -0.28 (0.07)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI [-0.43 to -0.03], Standard Error of Mean 0.10

9. Secondary Outcome: Change in Fructosamine From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mmol/L | -20.4 (3.22) | -9.6 (3.17)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Final Values) = -10.8, 95% CI [-19.9 to -1.8], Standard Error of Mean 4.55

10. Secondary Outcome: Change in 2-hour Mean Weighted PPG (After the Standardized Breakfast Meal) From Baseline to Week 4
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
mg/dL | -49.5 (6.61) | -13.2 (6.46)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -36.3, 95% CI [-54.7 to -17.9], Standard Error of Mean 9.25

11. Secondary Outcome: Change in Static Insulin Secretion Rate (10^-9 Min^-1) From Baseline to Week 4 - ITT Population
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Error); unit: 10^-9 min^-1
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 50
10^-9 min^-1 | 8.4 (2.07) | 1.4 (1.98)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA; Mean Difference (Final Values) = 7.0, 95% CI [1.3 to 12.7], Standard Error of Mean 2.86

ADVERSE EVENTS:
Arm/Group | Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 3/50 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=50) | Placebo (N=50)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution & PI agree they will not use or disclose and confidential information to third parties for a period of 10 years from receipt